CLINICAL TRIAL: NCT03261505
Title: Mechanistic Studies on Video-guided Acupuncture Imagery Treatment of Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jian Kong, Assistant Professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 2017P000820
Record Dates: First submitted 2017-08-22; First posted 2017-08-25 (Actual); Results first posted 2025-11-05 (Actual); Last update posted 2025-11-05 (Actual); Status verified 2025-10

CONDITIONS: Osteoarthritis, Knee
Keywords: fMRI; acupuncture; osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Acupuncture Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- VGAIT (Experimental)
  Interventions: Device: Acupuncture
- VGAIT Control (Sham Comparator)
  Interventions: Device: Acupuncture
- Real Acupuncture (Active Comparator)
  Interventions: Device: Acupuncture
- Sham Acupuncture (Placebo Comparator)
  Interventions: Device: Acupuncture

INTERVENTIONS:
Device: Acupuncture — Patients will watch a video of themselves receiving acupuncture or a control video or receive real or sham acupuncture treatment.
  Other Names: Video of Acupuncture

SUMMARY:
The aim of this study is to investigate brain response and connectivity changes evoked by video-guided acupuncture imagery treatment (VGAIT) and verum and sham acupuncture in knee osteoarthritis patients to elucidate the underlying brain mechanisms of mind-body interaction, imagery, and acupuncture.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Knee osteoarthritis patients
* Ages 40 to 70 years old

Exclusion Criteria:

* Any contraindications to MRI scanning (claustrophobia, metal implants)
* Current or past history of major medical, neurological, or psychiatric illness other than knee osteoarthritis (including high blood pressure, heart disorders, impaired elimination, stomach problems, major kidney or liver problems, bleeding problems, severe dehydration, history of diabetes, history of asthma or other respiratory condition)
* Pregnancy
* Non fluent English speaker

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2019-08-04 (Actual); Primary Completion 2023-08-29 (Actual); Study Completion 2023-08-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Athinoula A. Martinos Center for Biomedical Imaging, Charlestown, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VGAIT | VGAIT Control | Real Acupuncture | Sham Acupuncture
Started | 30 | 30 | 34 | 31
Completed | 27 | 27 | 27 | 28
Not Completed | 3 | 3 | 7 | 3
Not completed — Withdrawal by Subject | 2 | 3 | 4 | 3
Not completed — unrelated surgery preventing the subject participating the study | 0 | 0 | 1 | 0
Not completed — Claustrophobic or can not provide proof of diagnosis | 0 | 0 | 2 | 0
Not completed — the subject can not concentrate to complete the questionnaire | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VGAIT | VGAIT Control | Real Acupuncture | Sham Acupuncture | Total
Number analyzed (Participants) | 30 | 30 | 34 | 31 | 125
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 19 | 24 | 24 | 22 | 89
  >=65 years | 11 | 6 | 10 | 9 | 36
Age, Continuous [Mean (Standard Deviation); unit: year] | 61.5 (8.2) | 59.7 (7.8) | 59.7 (7.6) | 61.6 (7.4) | 60.6 (7.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 20 | 22 | 20 | 79
  Male | 13 | 10 | 12 | 11 | 46
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 0 | 1
  Asian | 1 | 2 | 0 | 1 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 3 | 1 | 5 | 3 | 12
  White | 26 | 27 | 27 | 26 | 106
  More than one race | 0 | 0 | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 30 | 30 | 34 | 31 | 125

OUTCOME MEASURES:

1. Primary Outcome: fMRI Signal Increases
Description: fMRI measures changes in brain activity by detecting fluctuations in blood oxygenation levels. The primary signal used in fMRI is the Blood Oxygen Level Dependent (BOLD) signal, which reflects neuronal activity indirectly through hemodynamic responses.
Time Frame: Collected once during the first treatment session
Population: SPM 12 was applied to investigate the brain responses to different interactions. Group analysis was performed using a random-effects model. A one-sample t-test was performed to compare the fMRI signal changes during manipulation vs. no manipulation within each treatment. Thresholds of p < 0.005 were applied. Peak values of fMRI signal increase brain regions (insula) were used for the report below.
Measure: Mean (Standard Deviation); unit: beta value of bold signal
Arm/Group | VGAIT | VGAIT Control | Real Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 23 | 26 | 24 | 25
beta value of bold signal | .42 (.27) | .48 (.47) | .47 (.37) | .33 (.32)

2. Secondary Outcome: PAG Resting State Connectivity
Description: The resting state functional connectivity of periaqueduct grey (PAG) before and after intervention. Resting-state functional connectivity (rsFC) is assessed by analyzing spontaneous BOLD signal fluctuations in different brain regions when a subject is at rest, providing insights into intrinsic brain network organization. Preprocessing steps, including motion correction, spatial normalization, and noise removal, ensure data accuracy.
Time Frame: baseline and after one month treatment
Population: The functional connectivity analysis was performed using CONN toolbox. A threshold of p < 0.005 was applied. We used peak brain regions showing significant functional connectivity increases after interventions to report (i.e. for VGAIT, insula was used; for VGAIT control, hippocampus was used; for verum acupuncture, insula was used; for sham acupuncture, prefrontal cortex was used). Please note this is NOT a result, rather a description on analysis details.
Measure: Mean (Standard Deviation); unit: normalized correlation coefficient
Arm/Group | VGAIT | VGAIT Control | Real Acupuncture | Sham Acupuncture
Number analyzed (Participants) | 22 | 25 | 21 | 25
normalized correlation coefficient | .09 (.13) | .09 (.1) | .1 (.08) | .08 (.12)

ADVERSE EVENTS:
Time Frame: Through the whole interventions, average about one month.
Arm/Group | VGAIT | VGAIT Control | Real Acupuncture | Sham Acupuncture
All-Cause Mortality (participants affected / at risk) | 0/30 | 0/30 | 0/34 | 0/31
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 0/34 | 0/31
Other Adverse Events (participants affected / at risk) | 0/30 | 0/30 | 1/34 | 0/31
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VGAIT (N=30) | VGAIT Control (N=30) | Real Acupuncture (N=34) | Sham Acupuncture (N=31)
Ringing of ear (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) — The subject experienced ear ring after MRI. It is not related to acupuncture treatment as the subject did not receive acupuncture treatment yet. The subject recovered without treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-02-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT03261505/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-08): https://cdn.clinicaltrials.gov/large-docs/05/NCT03261505/SAP_001.pdf